CLINICAL TRIAL: NCT01847599
Title: Implementation of a Therapeutic Educational Program Applicated to Adherence of Patients Treated by Capecitabine Alone or in Combination With Lapatinib
Brief Title: Educational Intervention to Adherence of Patients Treated by Capecitabine +/- Lapatinib
Acronym: ProMETheX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis : discontinuation for efficacy of the intervention
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A01300-39
Record Dates: First submitted 2013-04-05; First posted 2013-05-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Breast Cancer; Colorectal Cancer
Keywords: educational intervention; adherence; capecitabine; lapatinib
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- capecitabine (Other): patients treated by capecitabine alone (n=100)
  Interventions: Other: Educational Intervention to enhance the adherence of Patient treated by capecitabine +/- Lapatinib
- capecitabine + lapatinib (Other): patients treated by capecitabine and lapatinib (n=100)
  Interventions: Other: Educational Intervention to enhance the adherence of Patient treated by capecitabine +/- Lapatinib

INTERVENTIONS:
Other: Educational Intervention to enhance the adherence of Patient treated by capecitabine +/- Lapatinib

SUMMARY:
The purpose of this study is to evaluate the efficacy of the implementation of an educational program on adherence to capecitabine alone or in combination to lapatinib.

DETAILED DESCRIPTION:
200 subjects who meet the inclusion/exclusion criteria treated by capecitabine +/- lapatinib, will be enrolled into the study. Adherence to treatment of all subjects will be assessed during a first adherence evaluation period of 3 cycles in order to identify patients who need educational intervention(non adherent patients). Only nonadherent patients (adherence rate < 80%) will receive an education intervention. During the educational program, the efficacy of the implementation of an educational program on adherence to capecitabine alone or in combination to lapatinib will be evaluated for the 6 subsequent cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* histologically confirmed breast cancer or colorectal cancer
* Patient starting oral treatment : capecitabine alone or in combination with lapatinib (can be included before the first cycle or during the first 2 cycles).
* Volunteer to participate in the study.
* ambulatory treated patient
* Able to read, write and understand French.
* Subject who accept to use MEMS monitors to automatically compile their drug dosing histories
* Written informed consent

Exclusion Criteria:

* more than 3 metastatic chemotherapies
* any severe concomitant condition which makes it undesirable for the patient to participate in the study or which would jeopardize adherence with trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-09-06 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2017-07-02 (Actual)

PRIMARY OUTCOMES:
evaluation of the efficacy of the implementation of an educational program on adherence to capecitabine alone or in combination to lapatinib | every visit during 3 cycles i.e. 9 weeks (adherent patients) and for 6 additional cycles i.e. 18 weeks during educational intervention (nonadhererent patients)
  the efficacy of the implementation of an educational program will be evaluated by adherence assessment using electronic monitoring system

SECONDARY OUTCOMES:
patient satisfaction to the educational program as determined by questionnaire | at the end of the educational program i.e. approximately during the week 27
safety and tolerability as determined by adverse events frequency | for 3 cycles e.i. 9 weeks (adherent patients) or 9 cycles e.i. 27 weeks (nonadherent patients)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle VAN PRAAGH, MD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France